CLINICAL TRIAL: NCT00899899
Title: A Study of the Mechanisms of Intrinsic and Acquired Methotrexate Resistance in Acute Lymphocytic Leukemia
Brief Title: Resistance to Methotrexate in Patients With Acute Lymphoblastic Leukemia in Relapse or Remission
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: B977; COG-B977 (Other: Children's Oncology Group); CDR0000078589 (Other: Clinical Trials.gov)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia
Keywords: adult acute lymphoblastic leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: microarray analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about cancer and the development of drug resistance in patients.

PURPOSE: This laboratory study is looking at resistance to methotrexate in patients with acute lymphoblastic leukemia in relapse or remission.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the mechanisms of intrinsic and acquired methotrexate resistance using in vitro assays of matched initial diagnosis, relapsed, and nonrelapsed (control) leukemic blast samples from patients with acute lymphoblastic leukemia in relapse or remission.
* Determine if the mechanisms of acquired methotrexate resistance are related to dosage or timing of methotrexate administration or other clinical factors in these patients.

OUTLINE: Random samples of frozen leukemic blasts from relapsing patients at initial diagnosis and relapse are selected. A corresponding sample from nonrelapsing patients (control) at initial diagnosis is also randomly selected.

Reduced folate carrier (RFC) and dehydrofolate reductase (DHFR) expression is measured using a quantitative reverse transcriptase-polymerase chain reaction assay of prepared RNA. DHFR gene amplification is measured by a dot blot analysis of prepared DNA. Results of these assays are used to determine if a particular mechanism of acquired methotrexate resistance is associated with a particular subset of acute lymphoblastic leukemia patients. Data are collected regarding the actual timing and dosage of methotrexate received by each patient and are correlated with the mechanisms of resistance.

PROJECTED ACCRUAL: A total of 135 paired samples will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Acute lymphoblastic leukemia (ALL) in relapse, including all risk groups and leukemia subtypes, with frozen leukemic blast samples stored from the time of initial diagnosis and relapse
  * Non-relapsing ALL (as control)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute lymphoblastic leukemia (ALL) in relapse
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 1998-06; Primary Completion 2005-03 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Mechanisms of intrinsic and acquired methotrexate resistance
Correlation of acquired methotrexate resistance with dosage or timing of methotrexate administration
Correlation of acquired methotrexate resistance with other clinical factors

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gorlick, MD, Study Chair — Children's Hospital at Montefiore